Document Date: May 24, 2019

## The Effect Of Preoperative Parameters On Success After Descemet Membrane Endothelial Keratoplasty (DMEK) Surgery

| _ | | | |
|-----|---|---|--------|
| г | 1 | + | $\sim$ |
| -12 | ď | u | _ |

## INFORMED CONSENT FORM

## Dear Volunteer,

On the front of the eye is a transparent layer called the cornea. In this layer, hereditary corneal diseases may lose their transparency if they develop edema after a certain age or after cataract surgery. This situation causes visual impairment. In these cases, translucent corneal tissue taken from another person can be transplanted, and this transplant is called keratoplasty. Keratoplasty surgery can be done with a full layer of the cornea or some layers of the cornea. Descemet Membrane Endothelial Keratoplasty (DMEK) is the process of replacing the lower layer of the cornea, which is only closer to the eye, but not the full layer. The back layer of the cornea, the endothelial layer, is transplanted. Air is introduced into the eye to facilitate the attachment of the donor tissue. This air is drawn slowly by itself within 1 week. DMEK is most commonly performed in permanent corneal edema, called bullous keratopathy.

Optical coherence tomography is the process of scanning various layers of the eye in cross-section with high resolution using low energy light rays. During the examination of DMEK surgeries, OCT images are taken during the examination. Specular microscopy is an examination method that counts the cells in the area of surgery. Corneal topography is the method that provides an examination of the corneal structure and refraction. Control of the operation area can be done with these examinations made in the cornea region.

In our study titled 'The effect of anterior segment parameters on surgical success in patients undergoing Descemet Membrane Endothelial Keratoplasty (DMEK)', films taken during routine examinations in bullous keratopathy patients who underwent DMEK surgery will be examined. If you continue regular controls, data will be taken from your file once. It is planned to include 60 cases with bullous keratopathy disease in the study.

When filling out these forms, you will be able to get help from the researcher doctors with any questions. You will not have any financial obligations under the research. As part of the research, you will not be asked for an additional examination (other than those required for your disease). In connection with the research, no changes will be made regarding the treatment of your disease. If you do not agree to participate in the research or give up afterward, there will be no change or disruption in your treatment, and you can refuse to participate in the research and withdraw from the research at any time without losing any right or penalty. Audiences, attendants, ethics committee, institution, and other relevant health authorities will have direct access to the volunteer's original medical records, but this information will be kept confidential and will be granted by the volunteer by signing the written informed volunteer form. Your personal information (name, surname, etc.) will not be published anywhere.

I have read all the comments on the informed volunteer form. The written and verbal explanation about the research whose subject and purpose was mentioned above was made by the doctor named below. I know that I voluntarily participate in the research, I can leave the research with or without reason, whenever I want. I agree to participate in the study "The effect of anterior segment parameters on surgical success in patients undergoing Descemet Membrane Endothelial Keratoplasty (DMEK)" without any pressure or strain.

| Volunteer Name | Signature | Date |
|-----------------|-----------|------|
| Researcher Name | Signature | Date |